CLINICAL TRIAL: NCT05665725
Title: Phase I Study of Cytokine Release Syndrome Prophylaxis and Treatment With Siltuximab
Brief Title: Siltuximab for the Prevention of CAR T Cell Related Cytokine Release Syndrome in Patients With CD19 Positive Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Timothy Voorhees (Other)
Responsible Party: Sponsor-Investigator, Timothy Voorhees, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-22031; NCI-2022-10248 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (siltuximab, biospecimen) (Experimental): Patients receive siltuximab IV prior to CE19.CAR-T cell therapy and as clinically indicated on study. Patients undergo CT scan or PET scan throughout the trial. Patients also undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Siltuximab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Siltuximab — Given IV
  Other Names: Anti-IL-6 Chimeric Monoclonal Antibody; cCLB8; CNTO 328; CNTO-328; Sylvant

SUMMARY:
This phase I trial tests the safety and side effects of siltuximab in preventing CAR T cell therapy related cytokine release syndrome in patients with CD19 positive non-Hodgkin lymphoma. Several of the major complications of CD19 directed chimeric antigen receptor T-cell therapy (CD19.CAR-T) include cytokine release syndrome (CRS, a complication of a highly active immune system seen with some cancer treatments including CD19.CAR-T cell therapy) and immune effector cell therapy associated neurotoxicity (ICANS, neurologic complications related to an activated immune system seen with immunotherapy and CD19.CAR-T cell therapy). Siltuximab is a chimeric (having parts of different origins) murine (from mice) antibody that binds directly to IL-6 (a cytokine/ body chemical causing toxicities) and allows for its clearance. IL-6 is known to increase in a patient's blood after CD19.CAR-T cell infusion and has been associated with development of CRS and ICANS. Giving siltuximab prior to CD19.CAR-T cell therapy may help reduce CRS and/or ICANS after therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of siltuximab when given prior to CD19.CAR-T cells for prevention of cytokine release syndrome associated CAR-T cell therapy.

SECONDARY OBJECTIVES:

I. To describe the safety profile of siltuximab as first line treatment of new onset grade >= 2 cytokine release syndrome (CRS).

II. To estimate the incidence of all-grade CRS and grade >= 3 CRS after CAR-T cell therapy with siltuximab prophylaxis.

III. To estimate the incidence of all grade immune effector cell associated neurotoxicity syndrome (ICANS) and grade >= 3 ICANS after CAR-T cell therapy with siltuximab prophylaxis.

IV. To describe the response rates of grade >= 2 CRS to treatment with a second dose of siltuximab.

V. To describe the disease response rates of lymphoma patients after CD19.CAR-T cell therapy with siltuximab prophylaxis.

VI. To estimate the progression free survival (PFS) in subjects treated with CD19.CAR-T cell therapy with siltuximab prophylaxis.

VII. To estimate the overall survival (OS) in subjects treated with CD19.CAR-T cell therapy with siltuximab prophylaxis.

EXPLORATORY OBJECTIVES:

I. To describe CD19.CAR-T cell expansion and persistence following treatment with siltuximab prophylaxis.

II. To describe changes in plasma cytokine concentrations in patients treated with CD19.CAR-T cells with prophylactic siltuximab.

III. To describe changes in peripheral blood immunophenotypes in patients treated with CD19.CAR-T cells with prophylactic siltuximab.

IV. To examine the role of complement activation on development and persistence of ICANS.

V. To examine the correlation between apheresis product, infusional CAR-T product, and pre-lymphodepletion immunophenotypes with CRS/ICANS and CD19.CAR- T clinical response.

OUTLINE:

Patients receive siltuximab intravenously (IV) prior to CE19.CAR-T cell therapy and as clinically indicated on study. Patients undergo computed tomography (CT) scan or positron emission tomography (PET) scan throughout the trial. Patients also undergo blood sample collection during screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information
* Age >= 18 years at the time of consent
* Diagnosis of non-Hodgkin lymphoma
* Eligible for standard of care CD19.CAR-T cell therapy including axicabtagene ciloleucel, tisagenlecleucel, brexucabtagene autoleucel and lisocabtagene maraleucel)
* Subjects with hepatitis B virus (HBV) can be included if on suppressive antiviral therapy and have no detectable viral load
* Subjects with hepatitis C virus (HCV) can be included if HCV ribonucleic acid (RNA) viral load is undetected
* Measurable disease of > 1.5 cm in diameter and/or bone marrow involvement
* White blood cell count >= 1.0 x 10^9/L (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Hemoglobin >= 8.0 x 10^9/L (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Platelets >= 50 x 10^9/L (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Creatinine =< 2.0 x upper limit of normal (ULN) (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Bilirubin =< 2.0 × upper limit of normal (ULN). Subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level > 2.0 mg/dL if their conjugated bilirubin is =< 2.0 × ULN) (obtained within 14 days prior to initiating study treatment)
* Aspartate aminotransferase (AST) =< 3.0 × ULN (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Alanine aminotransferase (ALT) =< 3.0 × ULN (obtained within 14 days prior to initiating study treatment)

  * Note: Hematology and other lab parameters that are =< grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Females of childbearing potential must have a negative serum pregnancy test within 3 days prior to registration

  * NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months. Documentation of postmenopausal status must be provided
* Females of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 12 months after treatment the last dose of siltuximab. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method or an intrauterine device that meets < 1% failure rate for protection from pregnancy in the product label
* Male subjects with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 12 months after the last dose of siltuximab
* Subjects with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the experimental regimen are eligible for the trial
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee
* FOR SILTUXIMAB TREATMENT OF CRS/ICANS: Any subject with grade 1 ICANS lasting > 12 hours
* FOR SILTUXIMAB TREATMENT OF CRS/ICANS: Any subject with grade >= 2 CRS after CD19.CAR-T cell therapy
* FOR SILTUXIMAB TREATMENT OF CRS/ICANS: Any subject with grade >= 2 CRS after CD19.CAR-T cell therapy with concurrent ICANS
* SECOND SILTUXIMAB TREATMENT DOSE FOR CRS/ICANS: Subjects meeting criteria for a treatment dose who have received a treatment dose and have no change in the CRS or ICANS grade after 12 hours

Exclusion Criteria:

* Subjects requiring daily corticosteroids at a dose > 10mg of prednisone per day (orequivalent). Pulsed steroids for disease control are acceptable
* Subjects who are planned to receive prophylactic steroids for mitigating CRS/ICANS before, during, or after CD19.CAR-T infusion
* Active central nervous system or meningeal involvement by lymphoma. Subjects with symptoms of possible central nervous system (CNS) disease should undergo CNS workup with magnetic resonance imaging (MRI) brain and diagnostic lumbar puncture prior to enrollment on this study. Subjects with a history of CNS or meningeal involvement must be in a documented remission by cerebrospinal spinal fluid (CSF) evaluation and contrast-enhanced MRI imaging for at least 90 days prior to registration
* Patients with history of clinically relevant and active CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease
* Human immunodeficiency virus (HIV) seropositivity
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study and lactating females must agree to not breastfeed while taking study drugs)
* Uncontrolled concomitant illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association (NYHA) Class III or IV), unstable angina pectoris, myocardial infarction within 1 month prior to enrollment, uncontrolled cardiac arrhythmias, uncontrolled seizures, or severe non compensated hypertension (systolic blood pressure >= 180mmHg or diastolic blood pressure >= 120mmHg)
* FOR SILTUXIMAB TREATMENT OF CRS/ICANS: Subjects with CRS and no evidence of ICANS who require dexamethasone (or any steroid) due to severity of CRS as determined by the investigators
* FOR SILTUXIMAB TREATMENT OF CRS/ICANS: Prior history of a dose limiting toxicity (see section 6.5) due to siltuximab infusion according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) criteria v5.0
* SECOND SILTUXIMAB TREATMENT DOSE FOR CRS/ICANS: Subjects with CRS and no evidence of ICANS who require dexamethasone (or any steroid) due to severity of CRS as determined by the investigators
* SECOND SILTUXIMAB TREATMENT DOSE FOR CRS/ICANS: Prior history of a dose limiting toxicity due to siltuximab infusion according to NCI-CTCAE criteria v5.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Frequency and nature of adverse events associated with siltuximab prophylaxis prior to CD19 directed chimeric antigen receptor T-cell therapy (CD19.CAR-T) cell therapy | Up to 30 days after the last infusion of siltuximab
  Adverse events (AEs) will be described and classified per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 guidelines. The maximum grade of each type of toxicity will be extracted for each patient, and frequency counts will be tabulated to determine toxicity patterns, especially for grade 3 or above adverse events. The AE data associated with prophylaxis will be summarize for every patient: for patients receiving siltuximab only as prophylaxis, all AEs occur during the 30-day dose limiting toxicity observation period will be considered; for patients receiving siltuximab both as prophylaxis and as treatment, only the AEs occur before the treatment start will be considered for the primary endpoint.

SECONDARY OUTCOMES:
Frequency and nature of adverse events associated with siltuximab treatment of cytokine release syndrome (CRS) and/or immune effector cell associated neurotoxicity syndrome (ICANS) | Up to 30 days after the last infusion of siltuximab
  AEs will be described and classified per the NCI CTCAE v5.0 guidelines. The maximum grade of each type of toxicity will be extracted for each patient, and frequency counts will be tabulated to determine toxicity patterns, especially for grade 3 or above adverse events. AEs post treatment start will be summarized for the secondary endpoint.
Incidence of all grade CRS and grade >= 3 CRS | Up to 30 days after the last infusion of siltuximab
  According to American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading criteria.
Incidence of all grade ICANS and grade >= 3 ICANS | Up to 30 days after the last infusion of siltuximab
  According to ASTCT consensus grading criteria.
Percentage of participants who achieve resolution of CRS | At 24 hours from treatment
  Defined as absence of symptoms leading to diagnosis of CRS.
Objective response rate (complete response [CR] + partial response [PR]) | At day 30 following CD19.CAR-T cell therapy
  The ORR (CR + PR) will be calculated at the initial 30 day imaging assessment and 95% confidence interval computed.
Progression free survival | From the date of treatment initiation to date of progression or death, whichever occurs first, assessed up to 1 year
  Will be estimated using the Kaplan-Meier method.
Overall survival | From date of treatment initiation to date of death due to all causes, assessed up to 1 year
  Will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Voorhees, MD, MSCR, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT05665725/ICF_000.pdf